CLINICAL TRIAL: NCT01607034
Title: An Open-Label, Randomized, Crossover Study to Assess the Bioavailability of Dexpramipexole Administered in Soft Food and Water, and in Intact Tablet Form in the Fasted and Fed States in Healthy Volunteers
Brief Title: Study in Healthy Volunteers of the Bioavailability of Dexpramipexole Tablets and Food Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 223HV106
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 - tablet-fast (Experimental): 150 mg Dexpramipexole (intact tablet) single dose under fasted condition
  Interventions: Drug: Dexpramipexole
- Sequence 2 - tablet-fed (Experimental): 150 mg Dexpramipexole (intact tablet) single dose under fed condition
  Interventions: Drug: Dexpramipexole
- Sequence 3 - water-fast (Experimental): 150 mg Dexpramipexole single dose dispersed in water under fasted condition
  Interventions: Drug: Dexpramipexole
- Sequence 4 - apple-fast (Experimental): 150 mg Dexpramipexole single dose crushed and mixed in applesauce under fasted condition
  Interventions: Drug: Dexpramipexole

INTERVENTIONS:
Drug: Dexpramipexole — 150 mg single dose

SUMMARY:
To assess the bioavailability of dexpramipexole when mixed in soft food and water, and in intact tablet form in the fasted and fed states in healthy volunteers.

DETAILED DESCRIPTION:
The effect of food on dexpramipexole bioavailability following administration of the proposed commercial formulation (capsule-shaped tablet) at the anticipated therapeutic dose (150 mg twice daily) has not been studied. Therefore, this study has been designed to evaluate the effect of a standard high-fat, high-calorie meal on dexpramipexole bioavailability following administration of a single 150 mg dose in healthy volunteers, consistent with US Food and Drug Administration (FDA) and European Medicines Agency (EMA) recommendations.

Additionally, patients with ALS can have difficulty swallowing tablets, necessitating alternative methods of administration for the drug. Therefore, this study has also been designed to evaluate the bioavailability of dexpramipexole mixed with water or crushed in soft food (applesauce).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the Investigator, are healthy as determined by pre-study medical history, physical examination and 12-lead ECG.
* Adult males/females aged 18 to 55 years inclusive.
* Male subjects and female subjects of childbearing potential must practice effective contraception during the study and 90 days after their last dose of study drug.

Exclusion Criteria:

* History of malignant disease, including solid tumors and hematologic malignancies.
* History of any clinically significant endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major diseases, as determined by the Investigator.
* Surgery within 90 days prior to check in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
PK parameters of dexpramipexole including maximum plasma concentration (Cmax) and the area under the plasma concentration-time curve over time from 0 to infinity (AUC0-inf) of dexpramipexole. | zero to 48 hours post-dose

SECONDARY OUTCOMES:
Time to the maximum plasma concentration (Tmax), the area under the plasma concentration-time curve over time from 0 to t (AUC0-t) and terminal half-life (t½) of dexpramipexole. | zero to 48 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Saint Paul, Minnesota, United States